CLINICAL TRIAL: NCT04516031
Title: Posterior Component Separation With Transversus Abdominis Muscle Release Versus Mesh Only Repair in the Treatment of Complex Ventral Wall Hernia: A Randomized Controlled Trial
Brief Title: Transversus Abdominis Muscle Release Versus Mesh Only Repair in the Treatment of Complex Ventral Wall Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Co-supervisor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Transversus Abdominis Release
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Hernia, Ventral; Hernia Incisional; Hernia, Abdominal
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia; Hernia, Abdominal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesh-only repair (Active Comparator)
  Interventions: Procedure: Mesh-only repair
- Transversus Abdominis Muscl (Active Comparator)
  Interventions: Procedure: Posterior Component Separation with Transversus Abdominis Muscle Release

INTERVENTIONS:
Procedure: Posterior Component Separation with Transversus Abdominis Muscle Release — The posterior component separation technique with transversus abdominis muscle release was done as prescribed in Novitsky et al in 2012.
  Other Names: Transversus Abdominis Muscle Release
  Arms: Transversus Abdominis Muscl
Procedure: Mesh-only repair — The prosthetic mesh only repair was done as described by Wantz in 1991.
  Arms: Mesh-only repair

SUMMARY:
This trial was designed as a prospective randomized, controlled, intervention, with two parallel groups, and a primary endpoint of recurrence during 12 months' follow-up after initial treatment, with the randomization, was performed by an online software a 1:1 allocation.

DETAILED DESCRIPTION:
Eligibility Criteria

* both sexes
* aged between 18 and 65 years old
* presented complex ventral wall hernia or incisional hernia

Exclusion

* pregnant
* patients on steroid therapy
* underwent their hernia repair on an emergency basis

Interventions

* Eligible patients were randomized in equal proportions between "Mesh Only Repair" and "Posterior Component Separation with Transversus Abdominis Muscle Release"

ELIGIBILITY:
Inclusion Criteria:

* patients with complex ventral-wall and incisional hernia

Exclusion Criteria:

* pregnant female
* steroid therapy
* emergency basis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | after 12 months
  Reappearance of symptoms or swelling

SECONDARY OUTCOMES:
Morbidity | 30 days postoperative
  postoperative morbidity
Mortality | 30 days postoperative
  Postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shalaby, MD, MSc, PhD, Study Director — Mansoura University
Locations (1):
- Faculty of Medicine Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rabie M, Abdelnaby M, Morshed M, Shalaby M. Posterior component separation with transversus abdominis muscle release versus mesh-only repair in the treatment of complex ventral-wall hernia: a randomized controlled trial. BMC Surg. 2022 Sep 20;22(1):346. doi: 10.1186/s12893-022-01794-7. PMID 36127722